CLINICAL TRIAL: NCT05770739
Title: Application of Enhanced Recovery After Surgery During the Perioperative Period in Infants With Choledochal Cyst- a Multi-center Randomized Clinical Trial
Brief Title: A RCT Study of ERAS in Infants With Choledochal Cyst
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Children's Hospital (Other)
Responsible Party: Principal Investigator, Weibing Tang, professor, Nanjing Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 202204038-1
Record Dates: First submitted 2023-01-30; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-02

CONDITIONS: Enhanced Recovery After Surgery; Infant ALL; Cholangiectasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS group (Other): To apply accelerated rehabilitation surgery to children with biliary dilatation during perioperative period
  Interventions: Behavioral: Perioperative accelerated rehabilitation surgical measures
- placebo group (Other): In this gruop,Children with cholangiectasia were given traditional perioperative treatment
  Interventions: Behavioral: Traditional treatment

INTERVENTIONS:
Behavioral: Perioperative accelerated rehabilitation surgical measures — To apply accelerated rehabilitation surgery to children with biliary dilatation during perioperative period
  Arms: ERAS group
Behavioral: Traditional treatment — To provide traditional perioperative treatment for children with cholangiectasia
  Arms: placebo group

SUMMARY:
Recently, with reference to the successful experience of accelerated rehabilitation surgery in the field of adult surgery, the investigators have conducted studies on ERAS in pediatric and even infant cholangiectasia surgery to discuss its feasibility and safety. The results showed that some items of ERAS could be safely applied in perioperative management of CBD, and could reduce traumatic stress and promote postoperative recovery. Therefore, the investigators assumed that the ERAS protocols could be safely applied in the treatment of CBD in children and even infants, reducing traumatic stress in children with CBD, promoting postoperative rehabilitation, reducing complications and hospitalization time, reducing hospitalization costs, and saving medical resources.

DETAILED DESCRIPTION:
1. Optimize preoperative, intraoperative and postoperative perioperative management by learning from the successful experience of accelerated rehabilitation surgery model in other fields.

   For example: necessary and sufficient preoperative education of children and guardians; short fasting before surgery; oral carbohydrate at 2h before surgery; breast feeding at 4h before surgery (formula feeding at 6h before surgery); improved intestinal preparation; irregular placement of nasogastric tube; the use of general anesthesia plus epidural or sacral block anesthesia during surgery; attention to the whole process of heat preservation; strict control of infusion volume; and selection of minimally invasive hands Methods of operation; early postoperative activity, multi-mode analgesia, etc.
2. According to the pathophysiological characteristics of infants with cholangiectasia, several aspects were studied: minimally invasive surgery；promote gastrointestinal motor function recovery；develop principles and plans for early postoperative feeding；Rational placement of abdominal drainage tube; precise choice of anesthesia method, etc.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 0-12 months
* According to the clinical manifestations and preoperative imaging examination, the children admitted to hospital were diagnosed with choledochal cyst
* The legal guardian of the child signs the Informed Consent

Exclusion Criteria:

* Have potentially life-threatening diseases of various organ systems
* Preoperatively associated with other diseases that interfere with the treatment process of the child
* Caroli's disease was diagnosed
* Any other condition that the investigator deems unsuitable for participation in the trial

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
postoperative length of stay | through study completion, an average of 1 year
  To record the postoperative length of stay

SECONDARY OUTCOMES:
gastrointestinal functional recovery | through study completion, an average of 1 month
  To record the time of first exhaust and defecation and the time to return to full oral diet
Gastrointestinal decompression tube indwelling time | through study completion, an average of 1 month
  To calculate the indwelling time of Gastrointestinal decompression tube after surgery
Peritoneal drainage tube indwelling time | through study completion, an average of 1 month
  To calculate the indwelling time of Peritoneal drainage tube
Blood cortisol level | 24 hours after surgery
  To test the consentration of cortisol in blood
IL-6 level | 24 hours after surgery
  To test the consentration of IL-6 in blood
IL-10 level | 24 hours after surgery
  To test the consentration of IL-10 in blood
C-reactive protein (CRP) | 24 hours after surgery
  To test the consentration of CRP in blood
complication rate | one month after surgery
  to observe postoperative pulmonary infection, infection of incision, baby, abdominal cavity infection and the occurrence of complications such as anastomotic fistula, cholangitis.
Hospitalization expenses | through study completion, an average of 1 month
  the hospitalization cost of the child
Parents satisfaction score | through study completion, an average of 1 month
  To investigate the "Parents satisfaction score scale" (minimum=0, maximun=100); the higher scores mean a better outcome.
30-day readmission rate | one month after surgery
  To record the 30-day readmission rate after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Lv, Master, Principal Investigator — Children's Hospital of Nanjing Medical University
Locations (1):
- Children's Hospital of Nanjing Medical University, Nanjing, Jiangsu, China